CLINICAL TRIAL: NCT00490555
Title: The Effect of Male Hormonal Contraceptive Regimens on Prostate Tissue In Normal Men
Brief Title: PROS-1-Male Hormonal Contraceptive Regimens on Prostate Tissue
Acronym: PROS-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie T. Page, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31434-A; RFA-HD-06-014;; 06-4795-A 01 (Other: University of Washington IRB (old application number))
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Male Contraception; Testosterone; Testis; Contraception; Prostate
MeSH Terms: interventions — Testosterone; Dutasteride; N,N-dimethyl-4-anisidine; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): Placebo gel + Placebo pill + placebo injection
  Interventions: Other: Placebo Testosterone gel; Other: Placebo dutasteride; Other: Placebo DMPA
- 2 (Active Comparator): Testosterone 1% transdermal gel 10 g + placebo pill + placebo injection
  Interventions: Drug: Testosterone gel
- 3 (Active Comparator): Testosterone 1% transdermal gel 10 g + dutasteride 0.5 mg Orally + placebo injection
  Interventions: Drug: Testosterone gel; Drug: Dutasteride
- 4 (Active Comparator): Testosterone 1% transdermal gel 10 g + placebo pill + DMPA 300 mg injection (IM)
  Interventions: Drug: Testosterone gel; Drug: Depo-Medroxyprogesterone (DMPA); Other: Placebo dutasteride

INTERVENTIONS:
Drug: Testosterone gel — Testosterone gel 10 g
  Other Names: Testim
  Arms: 2; 3; 4
Drug: Dutasteride — dutasteride 0.5 mg orally
  Other Names: Avodart
  Arms: 3
Drug: Depo-Medroxyprogesterone (DMPA) — 300 mg DMPA injection on Day 0 IM (into the muscle)
  Other Names: Depo-Provera
  Arms: 4
Other: Placebo Testosterone gel — Place gel applied daily for 12 weeks
  Arms: 1
Other: Placebo dutasteride — placebo pill for 12 weeks
  Arms: 1; 4
Other: Placebo DMPA — placebo DMPA injection Once
  Arms: 1

SUMMARY:
The investigators propose to examine the in vivo responses to hormonal manipulation at the molecular level directly in the tissue of interest (prostate). As in the investigators' previous, pilot study, the investigators will use the novel approach of procuring tissue specimens from normal, healthy men who might be chose to use a male hormonal contraceptive regimen were it available. The investigators will employ state of the art techniques such as laser capture microdissection (LCM) and cDNA microarrays to determine the tissue-specific consequences of male hormonal contraceptive regimens on the prostate. The results will help guide the design, safety monitoring, and selection of male hormonal contraceptive agents and provide valuable insights into prostate human prostate biology.

The investigators will test the hypothesis that exogenous T administration that results in increased circulating T and dihydrotestosterone (DHT) levels will increase intraprostatic concentrations of T and its metabolite DHT.

The investigators will test the hypothesis that the addition of a potent 5α-reductase inhibitor, dutasteride, or the progestin, Depomedoxyprogesterone (IM DMPA), to T administration in young and middle aged men will decrease intraprostatic DHT and increase intraprostatic T concentrations compared to T alone.

The investigators will test the hypothesis that the addition of a 5α-reductase inhibitor dutasteride or the progestin IM DMPA to exogenous T, by reducing intraprostatic DHT, will decrease prostate epithelial proliferation, assessed by Ki-67 labeling index (Ki-67LI), and increase apoptosis, assessed by caspase-3 expression, and decrease androgen-regulated protein expression such as prostate specific antigen (PSA).

The investigators will test the hypothesis that the addition of a 5α-reductase inhibitor or the progestin IM DMPA to exogenous T, by modifying the intraprostatic hormonal milieu, will alter prostate epithelial gene expression. Specifically, the investigators expect that the addition of the 5α-reductase inhibitor dutasteride or the progestin IM DMPA to exogenous T, will result in decreased expression of androgen-regulated genes such as PSA.

DETAILED DESCRIPTION:
The purpose of this research study is to understand the effects of testosterone on the prostate. This knowledge will be used to help in the development of a safe male hormonal contraception.

We will be administering three drugs in this study: Testim (testosterone (T) gel), dutasteride (which affects testosterone break down) and Depomedoxyprogesterone (DMPA, a progestin). We want to see their effects on levels of hormones in the blood and prostate. In addition, we will be examining the effects of these drugs on the expression of genes within the prostate. DMPA suppresses LH and FSH, which are hormones made by the pituitary gland, thus blocking the signal from the brain that causes the testes to make testosterone. Prolonged (> 1 month) low levels of LH and FSH cause decreased sperm production in normal men. However, men may experience some side effects from the low levels of testosterone caused by DMPA; adding testosterone to DMPA eliminates these side effects while more effectively blocking LH and FSH release and sperm production. This combination of drugs is a promising male contraceptive regimen. However, the effect of these drugs on the prostate is not known. Some studies suggest that testosterone administration may promote prostate growth. Dutasteride blocks the conversion of testosterone to dihydrotestosterone and is used to treat men with enlarged prostates. Dutasteride shrinks the prostate. It is possible that combining testosterone and dutasteride may be an effective part of a male hormonal contraceptive regime. Therefore, further studies examining the effect of testosterone, DMPA and dutasteride on the prostate are needed.

ELIGIBILITY:
Inclusion Criteria:

* Men in good health, and without a history of chronic androgen therapy or known history of gonadal or prostate abnormalities.

  * PSA ≤ 2.
  * Age 25-55 years
  * Ability to understand the study,study procedures and provide consent
  * Normal serum total T, LH, FSH, urine analyses, and sperm count > or equal to 15million/ml
  * International Prostate Symptom Score (IPSS) < 10
  * Normal seminal fluid analysis (>20 million sperm/ml)
  * Agree not to donate blood during the treatment and recovery periods

Exclusion Criteria:

* A history or evidence of prostate or breast cancer
* History of invasive therapy for BPH
* History of acute urinary retention
* Current or past treatment with a 5α-reductase inhibitor
* History of anti/androgenic drugs or drugs that interfere with steroid metabolism within past 3 months
* Severe systemic illness (renal, liver, cardiac, lung disease, cancer, poorly controlled diabetes)
* Known untreated obstructive sleep apnea
* Hematocrit > 52%
* Skin disease that might interfere with T gel absorption
* Hypersensitivity to any of the drugs used in the study
* History of a bleeding disorder or anticoagulation
* History of drug or alcohol abuse within 12 months
* History of infertility or desire for fertility within 12 months, or current pregnant partner
* A first-degree relative (i.e. father, brother) with a history of prostate cancer
* Abnormal digital rectal examination or prostate ultrasound

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Page, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Amory JK, Page ST, Bremner WJ. Drug insight: Recent advances in male hormonal contraception. Nat Clin Pract Endocrinol Metab. 2006 Jan;2(1):32-41. doi: 10.1038/ncpendmet0069. PMID 16932251
- [Background] Brady BM, Amory JK, Perheentupa A, Zitzmann M, Hay CJ, Apter D, Anderson RA, Bremner WJ, Pollanen P, Nieschlag E, Wu FC, Kersemaekers WM. A multicentre study investigating subcutaneous etonogestrel implants with injectable testosterone decanoate as a potential long-acting male contraceptive. Hum Reprod. 2006 Jan;21(1):285-94. doi: 10.1093/humrep/dei300. Epub 2005 Sep 19. PMID 16172147
- [Background] Burkman R, Schlesselman JJ, Zieman M. Safety concerns and health benefits associated with oral contraception. Am J Obstet Gynecol. 2004 Apr;190(4 Suppl):S5-22. doi: 10.1016/j.ajog.2004.01.061. PMID 15105794
- [Background] Jacobsen SJ, Girman CJ, Lieber MM. Natural history of benign prostatic hyperplasia. Urology. 2001 Dec;58(6 Suppl 1):5-16; discussion 16. doi: 10.1016/s0090-4295(01)01298-5. PMID 11750242
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Wilson JD, George FW. The Physiology of Reproduction. Raven Press, 1994
- [Background] Russell DW, Wilson JD. Steroid 5 alpha-reductase: two genes/two enzymes. Annu Rev Biochem. 1994;63:25-61. doi: 10.1146/annurev.bi.63.070194.000325. No abstract available. PMID 7979239
- [Background] Thompson IM, Goodman PJ, Tangen CM, Lucia MS, Miller GJ, Ford LG, Lieber MM, Cespedes RD, Atkins JN, Lippman SM, Carlin SM, Ryan A, Szczepanek CM, Crowley JJ, Coltman CA Jr. The influence of finasteride on the development of prostate cancer. N Engl J Med. 2003 Jul 17;349(3):215-24. doi: 10.1056/NEJMoa030660. Epub 2003 Jun 24. PMID 12824459
- [Background] Geller J. Effect of finasteride, a 5 alpha-reductase inhibitor on prostate tissue androgens and prostate-specific antigen. J Clin Endocrinol Metab. 1990 Dec;71(6):1552-5. doi: 10.1210/jcem-71-6-1552. PMID 1699965
- [Background] Geller J, Albert J. Effects of castration compared with total androgen blockade on tissue dihydrotestosterone (DHT) concentration in benign prostatic hyperplasia (BPH). Urol Res. 1987;15(3):151-3. doi: 10.1007/BF00254427. PMID 3629749
- [Background] Mohler JL, Gregory CW, Ford OH 3rd, Kim D, Weaver CM, Petrusz P, Wilson EM, French FS. The androgen axis in recurrent prostate cancer. Clin Cancer Res. 2004 Jan 15;10(2):440-8. doi: 10.1158/1078-0432.ccr-1146-03. PMID 14760063
- [Background] Forti G, Salerno R, Moneti G, Zoppi S, Fiorelli G, Marinoni T, Natali A, Costantini A, Serio M, Martini L, et al. Three-month treatment with a long-acting gonadotropin-releasing hormone agonist of patients with benign prostatic hyperplasia: effects on tissue androgen concentration, 5 alpha-reductase activity and androgen receptor content. J Clin Endocrinol Metab. 1989 Feb;68(2):461-8. doi: 10.1210/jcem-68-2-461. PMID 2465302
- [Background] Habib FK, Ross M, Tate R, Chisholm GD. Differential effect of finasteride on the tissue androgen concentrations in benign prostatic hyperplasia. Clin Endocrinol (Oxf). 1997 Feb;46(2):137-44. doi: 10.1046/j.1365-2265.1997.950908.x. PMID 9135694
- [Background] Page ST, Lin DW, Mostaghel EA, Hess DL, True LD, Amory JK, Nelson PS, Matsumoto AM, Bremner WJ. Persistent intraprostatic androgen concentrations after medical castration in healthy men. J Clin Endocrinol Metab. 2006 Oct;91(10):3850-6. doi: 10.1210/jc.2006-0968. Epub 2006 Aug 1. PMID 16882745
- [Background] Page ST, Amory JK, Anawalt BD, Irwig MS, Brockenbrough AT, Matsumoto AM, Bremner WJ. Testosterone gel combined with depomedroxyprogesterone acetate is an effective male hormonal contraceptive regimen and is not enhanced by the addition of a GnRH antagonist. J Clin Endocrinol Metab. 2006 Nov;91(11):4374-80. doi: 10.1210/jc.2006-1411. Epub 2006 Aug 29. PMID 16940442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male volunteers, 25-55 yr old, were recruited via advertisement: flyers on University campus and newspaper ads.
Groups:
- 1) Placebo: Placebo gel + Placebo pill + placebo DMPA
- 2) Testosterone (T) Gel: Testosterone 1% transdermal gel 10g (Testim)+ placebo pill, daily + placebo DMPA
- 3) T Gel+Dutasteride: Testosterone 1% transdermal gel 10g + dutasteride 0.5mg Orally + placebo DMPA
- 4) T Gel+DMPA: Testosterone 1% transdermal gel 10g, daily + placebo Dutasteride pill, daily + DMPA 300mg injection (IM)
Period: Overall Study
Arm/Group | 1) Placebo | 2) Testosterone (T) Gel | 3) T Gel+Dutasteride | 4) T Gel+DMPA
Started | 8 | 8 | 9 | 7
Completed | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 2 | 0
Not completed — noncompliant with drug administration | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1) Placebo: Placebo Testosterone gel + Placebo Dutasteride pill + placebo DMPA
- 2) Testosterone Gel: Testosterone 1% transdermal gel 10g + placebo Dutasteride + placebo DMPA
- 3) T Gel +Dutasteride: Testosterone 1% transdermal gel 10g + dutasteride 0.5mg Orally + placebo DMPA
- 4) T Gel+ DMPA: Testosterone 1% transdermal gel 10g + placebo Dutasteride + DMPA 300mg injection (IM)
- Total: Total of all reporting groups
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA | Total
Number analyzed (Participants) | 8 | 8 | 9 | 7 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 7 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (7.72) | 37 (6.19) | 37 (8.45) | 39 (10.11) | 39 (3.46)
Sex/Gender, Customized [Number; unit: participants] — Male population, per protocol
  participants
    Female | 0 | 0 | 0 | 0 | 0
    Male | 8 | 8 | 9 | 7 | 32
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 7 | 32
Luteinizing Hormone (LH) [Median (Inter-Quartile Range); unit: IU/liter] | 4.0 [3.5 to 5.6] | 3.9 [2.7 to 5.5] | 5.3 [4.2 to 6.6] | 3.2 [2.7 to 4.0] | 4.1 [3.3 to 5.4]
Follical-stimulating hormone (FSH) [Median (Inter-Quartile Range); unit: IU/liter] | 3.6 [2.6 to 4.4] | 3.3 [2.6 to 3.7] | 4.0 [2.4 to 5.5] | 2.8 [2.6 to 4.2] | 3.4 [2.5 to 4.4]
SHBG [Median (Inter-Quartile Range); unit: nmol/liter] | 33 [24 to 45] | 36 [13 to 50] | 38 [26 to 52] | 33 [17 to 38] | 35 [20 to 46]
Testosterone (T) concentration [Median (Inter-Quartile Range); unit: ng/mL] | 3.9 [3.8 to 5.0] | 3.9 [2.9 to 5.9] | 4.8 [3.8 to 6.3] | 4.0 [3.0 to 5.8] | 4.1 [3.4 to 5.7]
Dihydrotestosterone (DHT) [Median (Inter-Quartile Range); unit: ng/mL] | 0.5 [0.4 to 0.5] | 0.6 [0.4 to 0.9] | 0.7 [0.6 to 1.0] | 0.6 [0.4 to 0.8] | 0.6 [0.4 to 0.8]
Prostate-Specific Antigen (PSA) [Median (Inter-Quartile Range); unit: ng/mL] | 0.7 [0.6 to 1.0] | 0.7 [0.4 to 1.1] | 0.9 [0.7 to 1.1] | 0.5 [0.4 to 0.6] | 0.7 [0.5 to 0.9]
Prostate volume [Median (Inter-Quartile Range); unit: ml] | 25 [16 to 29] | 15 [14 to 19] | 15 [13 to 21] | 19 [14 to 21] | 18 [14 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA)
Description: PSA level week 10 end of treatment
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Number analyzed (Participants) | 8 | 7 | 7 | 7
ng/mL | 0.8 [0.7 to 1.2] | 0.9 [0.3 to 1.2] | 0.7 [0.7 to 1.1] | 0.4 [0.4 to 0.6]

2. Primary Outcome: Testosterone Concentration
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Number analyzed (Participants) | 8 | 7 | 7 | 7
ng/mL | 4.0 [2.9 to 5.6] | 4.4 [3.2 to 6.2] | 7.0 [4.4 to 12.4] | 1.8 [1.3 to 2.9]

3. Primary Outcome: Dihydrotestosterone (DHT) Concentration
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Number analyzed (Participants) | 8 | 7 | 7 | 7
ng/mL | 0.5 [0.4 to 0.6] | 1.8 [1.2 to 2.5] | 0.5 [0.3 to 0.5] | 0.6 [0.2 to 1.8]

4. Secondary Outcome: Androstenedione (AED)
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Number analyzed (Participants) | 8 | 7 | 7 | 7
ng/mL | 0.9 [0.8 to 1.1] | 0.9 [0.8 to 1.3] | 1.8 [1.3 to 3.7] | 0.7 [0.6 to 1.0]

5. Secondary Outcome: Dehydroepiandrosterone (DHEA)
Time Frame: 10 weeks
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Number analyzed (Participants) | 8 | 7 | 7 | 7
ng/mL | 4.3 [2.7 to 5.5] | 3.5 [2.0 to 7.5] | 3.8 [3.8 to 6.3] | 3.2 [2.1 to 4.0]

ADVERSE EVENTS:
Arm/Group | 1) Placebo | 2) Testosterone Gel | 3) T Gel +Dutasteride | 4) T Gel+ DMPA
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 2/7 | 1/9 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1) Placebo (N=8) | 2) Testosterone Gel (N=7) | 3) T Gel +Dutasteride (N=9) | 4) T Gel+ DMPA (N=7)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — leg abscess - unrelated trauma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No